CLINICAL TRIAL: NCT01183507
Title: Task Specific Exercise for the Pre-Clinically Disabled
Brief Title: Task Specific Exercise for the Prevention of Disability
Acronym: TSE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 410-2009; 1R21AG031974-01A2 (NIH)
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Pre-Clinically Disabled

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NIA intervention (Active Comparator)
  Interventions: Behavioral: NIA intervention
- TSE intervention (Experimental)
  Interventions: Behavioral: TSE

INTERVENTIONS:
Behavioral: NIA intervention — The NIA physical activity intervention is of moderate intensity and will consist of aerobic, strength, flexibility, and balance training, with a target duration of 120 minutes per week.
  Arms: NIA intervention
Behavioral: TSE — The TSE intervention is also of moderate intensity and target duration of 120 minutes per week and will consist of exercises that closely mimic functional tasks, such as vacuuming, stair ascent and descent, and lifting a weighted laundry basket.
  Arms: TSE intervention

SUMMARY:
The purpose of this research study is to evaluate the effect of two different exercise programs on physical function in men and women 60 years of age and older.

DETAILED DESCRIPTION:
Pre-clinical disability is an early warning system in the disablement process as it is characterized by selecting to perform everyday tasks less often and compensating for those tasks still being performed. This phase serves as an ideal target for preventative strategies because treatments can be designed for individuals on the verge of disability thus interrupting the occurrence of outright disability. One such strategy that optimizes the transfer of adaptations to real-life situations is task-specific exercise (TSE). This type of intervention holds promise to determine how pre-clinically disabled older adults might interrupt the disablement process and instead begin an enablement process and thus lead us to better interventions to treat and prevent disability from occurring. However, because of the complexity of the disablement process, it has been extremely challenging to objectively identify outcomes that represent changes in selection, optimization, and compensation of tasks (the SOC domains). The objective of the current application is first, to ask what are the short and long-term responses of TSE in the pre-clinically disabled older adults (aged 60+ years). Thirdly, we will shed exciting new light on whether TSE alters neuromechanical and psychological factors. We want to know this, in part, from a mechanistic perspective to gain insight into the processes by which TSE improves disablement outcomes. Also, this will help us to better understand how to enhance the TSE intervention to treat pre-clinically disabled patients. Thus, we offer two hypotheses: Hypothesis #1: TSE increases selection and optimization of everyday tasks, while reducing compensation to achieve task performance. Hypothesis #2. TSE mediates changes in SOC domains through both neuromechanical (decrease variability of movement and increase muscle work capacity) and psychological (increased confidence to perform tasks and increased executive function) properties. These data are expected to guide us in designing a randomized controlled trial that will test whether TSE in the pre-clinically disabled can reduce future incidence of outright disability.

ELIGIBILITY:
Inclusion Criteria:

* Age: 60+ years
* Self-report no difficulty walking ½ mile, climbing steps, stooping-crouching-kneeling, getting up off the floor, or lifting/carrying something as heavy as 10 lbs
* Modified the method of frequency of walking ½ mile, climbing steps, stooping-crouching-kneeling, getting up off the floor or lifting/carrying something as heavy as 10 lbs
* Observed use of 7 or more modifications plus a score of 2 or greater on at least two tasks on the MOD scale
* Sedentary lifestyle ( < 125 minutes walking or performing aerobic exercise)
* Successful completion of the behavioral run-in without the assistance of a spouse or other family or friend
* Willing and able to participate in all aspects of the pilot study, i.e., randomization, pre- and post-testing, home evaluation
* Willing to give and informed consent

Exclusion Criteria:

* Self-reporting having "any difficulty" walking ½ mile, climbing steps, stooping-crouching-kneeling, getting up off the floor, or lifting/carrying something as heavy as 10 lbs
* Failure to give consent
* Active Treatment for cancer
* Stroke (<6 mo)
* Neurological disorder
* Peripheral vascular disease
* Congestive heart failure (NYHA class II, III or IV), coronary artery disease (myocardial infarction <6 mo) or valvular heart disease
* Major psychiatric disease
* Severe anemia
* Liver or renal disease
* Uncontrolled diabetes or hypertension
* Macular degeneration
* Blindness or deafness
* Orthopedic impairment
* Rheumatoid arthritis or severe osteoarthritis
* Fracture in upper or lower extremity within last 6 months
* Upper or lower extremity amputation
* Participation in another intervention trial
* Inability to perform exercise due to severe physical disability
* MMSE < 24
* Plans to move within the next year

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2010-04; Primary Completion 2012-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
MOD Score | Screening, 6, 12, 24 weeks
  Number of modifications used by participants in the performance daily activities

SECONDARY OUTCOMES:
400 m walk | Baseline, 12, 24 wks
  The 400-m walk was chosen because, clinically, it has been proposed as a threshold of high level of performance and is strongly associated with measures of functional limitations, disability and mortality, and predicts future loss of ability to complete the walk. The ability to walk 400 meters has demonstrated excellent test-retest reliability (Kappa = 1.0), based on independent assessments completed 1-7 days apart among 60 physically impaired older persons.
Short Physical Performance Battery | Baseline, 12, 24 wks
  The SPPB, based on a timed short distance walk, repeated chair stands and balance test (as described by Guralnik et al.), will be used to demonstrate the physical function of older adults. Each of the 3 performance measures will be assigned a score ranging from 0 to 4.
Late Life Function and Disability Instrument | Baseline, 12, 24 wks
  The Late Life Function and Disability Instrument, developed by Dr. Jette et al., will be used to document disability status using a scale from 0 to 100, with higher scores indicating higher levels of function. The instrument includes 16 tasks representing a broad range of disability indicators that assesses both frequency of doing a task and perceived limitation, and was developed using more contemporary psychometric techniques (Rasch models). The scale has recently shown strong concurrent and predictive validity with physical performance.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Manini, PhD, Principal Investigator — University of Florida Department of Aging and Geriatric Research
Locations (2):
- United States (2):
  - UF Aging and Rehabilitation Research Center, Gainesville, Florida
  - UF Institute on Aging Health Promotion Center, Gainesville, Florida

REFERENCES:
- See also: UF Department of Aging — http://aging.ufl.edu/